CLINICAL TRIAL: NCT02513498
Title: Ixazomib for Treatment of Chronic Graft vs. Host Disease
Brief Title: Ixazomib Citrate in Treating Patients With Chronic Graft-versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9292; NCI-2015-00882 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16032; 9292 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib citrate) (Experimental): Patients receive ixazomib citrate PO once weekly on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response, partial response, or stable disease may receive an additional 6 courses of ixazomib citrate.
  Interventions: Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well ixazomib citrate works in treating patients with chronic graft-versus-host disease. Chronic graft-versus-host disease is a complication of a donor bone marrow or blood cell transplant, usually occurring more than three months after transplant, in which donor cells damage the host tissue. Ixazomib citrate may be an effective treatment for chronic graft-versus-host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the proportion of subjects with treatment failure by 6 months of ixazomib (ixazomib citrate) treatment for chronic graft-versus-host disease (GVHD).

SECONDARY OBJECTIVES:

I. Determine 3 month overall (complete + partial), and complete response rate.

II. Determine 6 month overall (complete + partial), and complete response rate.

III. Report overall survival, non-relapse mortality, primary malignancy relapse, failure-free survival, treatment success, and discontinuation of immune-suppressive therapy at 6 months and 1 year.

IV. Examine functional outcome (2-minute walk test) and patient-reported outcomes (Lee Chronic GVHD Symptom Scale, quality of life [Short Form Health Survey (SF)-36, Functional Assessment of Cancer Therapy Bone Marrow Transplant (FACT-BMT)], Human Activity Profile [HAP]) at study enrollment, 6 months, and 1 year.

V. Study biologic effects of proteasome inhibition.

OUTLINE:

Patients receive ixazomib citrate orally (PO) once weekly on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response, partial response, or stable disease may receive an additional 6 courses of ixazomib citrate.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence or exclusively non-heterosexual activity when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice two effective contraception measures during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence or exclusively non-heterosexual activity when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Patients must have a diagnosis of a chronic GVHD according to the National Institute of Health (NIH) Consensus Criteria
* Patients must have failed at least one prior line of systemic immune suppressive therapy for management of chronic GVHD
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 75,000/mm^3; platelet transfusions are not allowed within 3 days before study enrollment
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Calculated creatinine clearance >= 30 mL/min

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Major surgery within 14 days before enrollment

  * Does not include placement of venous access device, bone marrow biopsy, GVHD diagnostic biopsy, or other routine procedures in chronic GVHD or post-transplantation care
* Uncontrolled infection within 14 days before study enrollment

  * Infection treated with appropriate antimicrobial therapy and without signs of progression/treatment failure does not constitute an exclusion criterion
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months

  * Chronic hypertension on medical therapy does not constitute an exclusion criterion
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Non-hematologic malignancy within the past 2 years with the exception of:

  * Adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer
  * Carcinoma in situ of the cervix or breast
  * Prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels
  * Cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study
* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Treatment with non-Food and Drug Administration (FDA) approved drug within 21 days of start of this trial
* New systemic immune suppressive agent added for the treatment of chronic GVHD within 2 weeks prior to enrollment

  * Addition of a new systemic immune suppressive treatment simultaneously with ixazomib is also prohibited
* Evidence of recurrent or progressive underlying malignant disease
* Karnofsky performance status < 70%
* Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ixazomib Citrate)
Started | 50
Completed | 26
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [44 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 43
  More than one race | 1
  Unknown or Not Reported | 2
Primary Disease [Count of Participants; unit: Participants]
  Acute leukemia (ALL/AML) | 26
  Chronic leukemia (CML/CLL) | 6
  Lymphoma (NHL/HD) | 9
  Myeloma | 2
  MDS/Myeloproliferative neoplasm | 4
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: According to National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0
Time Frame: Up to 30 days following completion of study treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
participants
  Serious Adverse Events | 19
  Non-Serious Adverse Events | 18

2. Primary Outcome: Probability of Treatment Failure at 6 Months
Description: Kaplan-Meier estimate assessed at 6 months for probability of treatment failure, defined as addition of a line of systemic immune-suppressive therapy, recurrent malignancy, or death.
Time Frame: 6 months
Measure: Number; unit: Treatment failure probability
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
Treatment failure probability | .28

3. Secondary Outcome: Biologic Studies
Description: The biologic impact of proteasome inhibition in the treatment of chronic GVHD will be assessed.
Time Frame: Up to 6 months
Population: Response to study drug too minimal to justify time and expense to perform biologic studies.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Complete Response (CR) Rate
Description: Response will be determined by both clinician-defined, as well as separately calculated according to the proposed response definitions of the NIH Consensus Conference.
Time Frame: 6 months
Population: Participants who could be evaluated for response (not missing data)
Measure: Count of Participants; unit: Participants
Groups:
- Response Evaluated by MD; Response Evaluated by NIH: Participants who receive ixazomib citrate
Arm/Group | Response Evaluated by MD | Response Evaluated by NIH
Number analyzed (Participants) | 42 | 43
Participants
  Partial Response | 16 | 17
  Mixed Response | 4 | 10
  Unchanged | 9 | 4
  Progressive | 3 | 2
  Failed | 10 | 10

5. Secondary Outcome: Probability of Non-relapse Mortality at 1 Year
Description: Kaplan-Meier estimate assessed at 1 year for probability of non-relapse mortality, defined as death in the absence of primary malignancy relapse after transplant.
Time Frame: 1 year
Measure: Number; unit: non-relapse mortality probability
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
non-relapse mortality probability | 0.1

6. Secondary Outcome: Cumulative Incidence of Primary Malignancy Relapse
Description: Defined as hematologic relapse or any unplanned intervention to prevent progression of disease in patients with evidence (molecular, cytogenetic, flow cytometric, radiographic) of malignant disease after transplantation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
Participants | 1

7. Secondary Outcome: Probability of Failure-free Survival at 1 Year
Description: Kaplan-Meier estimate assessed at 1 year for failure-free survival, defined as the absence of death from any cause, relapse or addition of secondary immune suppressive agents.
Time Frame: 1 year
Measure: Number; unit: probability of failure-free survival
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
probability of failure-free survival | 0.57

8. Secondary Outcome: Incidence of Discontinuation of All Systemic Immune Suppressive Therapies
Description: The incidence of complete discontinuation of all systemic immune-suppressive therapies will be determined at 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
Participants | 0

9. Secondary Outcome: Overall Response Rate (ORR) (Complete Response + Partial Response)
Description: ORR at 6 months will be determined by both clinician-defined categories of complete response and partial response, as well as separately calculated according to the proposed response definitions of the NIH Consensus Conference.
Time Frame: 6 months
Population: Participants with missing response data are counted as failures; primarily missing due to failure to collect data in patients who stopped study drug but did not experience treatment failure.
Measure: Number; unit: participants
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
participants
  Physician impression ORR | 16
  NIH ORR | 17

10. Secondary Outcome: Probability of Overall Survival at 1 Year
Description: Kaplan-Meier estimate assessed at 1 year for overall survival, defined as absence of death from any cause.
Time Frame: 1 year
Measure: Number; unit: probability of overall survival
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
probability of overall survival | .9

11. Secondary Outcome: Treatment Success
Description: Treatment success will be estimated at 1 year with a composite outcome of complete resolution of all reversible chronic graft-versus-host disease (GVHD) manifestations, discontinuation of all systemic immune suppressive agents, and freedom from death or primary malignancy relapse after transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
Participants | 0

12. Secondary Outcome: Use of Additional Systemic Immune Suppressive Therapies
Description: Addition of therapy after ixazomib constitutes failure, could occur at any time from baseline to 12mo.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 50
Participants | 21

13. Secondary Outcome: Symptoms as Measured by Patient Self-report--Short Form-36 (SF-36)
Description: SF-36 subscales have min=0 and max=100; results given are actual scores at 12mo, with higher scores indicating higher quality of life.
Time Frame: 1 year
Population: 25 of 50 participants were evaluable at 12mo due to missing patient survey data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 25
units on a scale
  norm-based physical functioning | 44.4 [25.5 to 57]
  norm-based role-physical score | 37.3 [27.5 to 56.9]
  norm-based bodily pain score | 46.1 [29.2 to 62.1]
  norm-based general health score | 36.2 [25.8 to 57.7]
  norm-based vitality score | 49 [27.1 to 70.8]
  norm-based social functioning score | 51.4 [29.6 to 56.8]
  norm-based role-emotional score | 48.1 [28.7 to 55.9]
  norm-based mental health score | 52.8 [27.5 to 64.1]
  standardized physical component score | 39.7 [27.1 to 54.8]
  standardized mental component score | 53.8 [32.7 to 63]

14. Secondary Outcome: Symptoms as Measured by Patient Self-report--Functional Assessment of Chronic Illness Therapy (FACT)
Description: FACT-BMT subscales have various min/max, see below; results given are actual 12mo scores, with higher scores indicating better functioning.
  FACT physical well-being (0-28) FACT social/family well-being (0-28) FACT emotional well-being (0-24) FACT functional well-being (0-28) FACT Bone Marrow Transplant (BMT) subscale (0-40) FACT trial outcome index (0-96) FACT-General (G) (0-108) FACT-BMT total (0-148)
Time Frame: 1 year
Population: 25 of 50 participants were evaluable at 12mo due to missing patient survey data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 25
units on a scale
  physical well-being | 23 [7 to 28]
  social/family well-being | 23.7 [12 to 28]
  emotional well-being | 21 [10 to 24]
  functional well-being | 18 [5.8 to 28]
  BMT subscale | 32 [16 to 36]
  FACT-G | 84.7 [55.8 to 105]
  trial outcome index | 72 [38.8 to 89]
  FACT-BMT total | 114.1 [75 to 140]

15. Secondary Outcome: Symptoms as Measured by Patient Self-report--Human Activities Profile (HAP)
Description: HAP subscales have min=0 and max=94; results given are actual 12mo scores, with higher scores indicating better functioning.
  Maximum Activity Score (MAS) is highest item number answered still doing. Represents highest oxygen demanding activity that respondent still performs.
  Adjusted Activity Score (AAS) is MAS minus total number of stopped doing responses below MAS. A measure of usual daily activities.
  Modified AAS is MAS minus total number of stopped doing responses below MAS but not penalized for not doing activities not permitted post transplant. The following items are not counted against the score:11,15,19,20,22,25,34,41,42,47,49,50,52,53,54,57,72,73,77,78.
Time Frame: 1 year
Population: 25 of 50 participants were evaluable at 12mo due to missing patient survey data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 25
units on a scale
  maximum activity score | 74 [28 to 91]
  adjusted activity score | 70 [24 to 88]
  modified adjusted activity score | 70 [24 to 88]

16. Secondary Outcome: Symptoms as Measured by Patient Self-report--Lee Chronic GVHD Symptom Scale
Description: Lee symptom scale (LSS) has subscales with min=0, max=100; results given are 12mo scores, with higher numbers indicating higher symptom burden.
Time Frame: 1 year
Population: 25 of 50 participants were evaluable at 12mo due to missing patient survey data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Ixazomib Citrate)
Number analyzed (Participants) | 25
units on a scale
  skin scale | 15 [0 to 45]
  energy scale | 25 [0 to 87.5]
  lung scale | 10 [0 to 60]
  eye scale | 50 [0 to 100]
  nutrition scale | 0 [0 to 25]
  psychological scale | 16.7 [0 to 58.3]
  mouth scale | 0 [0 to 37.5]
  overall summary score | 20.8 [4.3 to 50]

ADVERSE EVENTS:
Time Frame: 30 days after stopping study drug
Arm/Group | Treatment (Ixazomib Citrate)
All-Cause Mortality (participants affected / at risk) | 5/50
Serious Adverse Events (participants affected / at risk) | 19/50
Other Adverse Events (participants affected / at risk) | 18/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate) (N=50)
Death (General disorders) | 1 (1) — Unknown cause
Calcaneal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
vomiting, nausea, diarrhea (Gastrointestinal disorders) | 1 (1)
chills/weakness (General disorders) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
right bundle branch block (Cardiac disorders) | 1 (1)
flu-like symptoms (General disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
skin infection (Infections and infestations) | 1 (1)
avascular necrosis of hip (Musculoskeletal and connective tissue disorders) | 1 (1)
perforated colon (Gastrointestinal disorders) | 1 (1)
periorbital cellulitis (Eye disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fever (General disorders) | 3 (4)
osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Progressive multifocal leukoencephalopathy (Nervous system disorders) | 1 (1)
leg ulcers/cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
pericardial effusion (Cardiac disorders) | 1 (1)
acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate) (N=50)
amylase increased (Investigations) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (3)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
influenza a (Infections and infestations) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
lipase increased (Investigations) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
peripheral neuropathy (Nervous system disorders) | 2 (2)
otomastoiditis (Ear and labyrinth disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
restlessness (Nervous system disorders) | 1 (1)
skin infection (Infections and infestations) | 1 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 3 (5)
worsening pain (Musculoskeletal and connective tissue disorders) | 1 (1)
wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02513498/Prot_SAP_000.pdf